CLINICAL TRIAL: NCT03627663
Title: Dialectic Behavior Treatment Skills System (DBT-SS) as Treatment for Cognitively Challenged Individuals With Deliberate Self-harm
Brief Title: DBT-SS for Cognitively Challenged Individuals With Deliberate Self-harm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Sofie Westling, Senior Psychiatrist, Doctor of Medicine, Region Skane
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017/827
Record Dates: First submitted 2017-12-21; First posted 2018-08-13 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-06

CONDITIONS: Self Harm; Suicide, Attempted; Borderline Personality Disorder
MeSH Terms: conditions — Self-Injurious Behavior; Suicide, Attempted; Borderline Personality Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Receiving treatment with Dialectic Behavior Therapy - Skills System + Treatment As Usual
  Interventions: Behavioral: Dialectic Behavior Therapy - Skills System

INTERVENTIONS:
Behavioral: Dialectic Behavior Therapy - Skills System — Treatment with Dialectical Behavior therapy adapted for cognitively challenged individuals

SUMMARY:
The study evaluates the effect of Dialectic Behavior Therapy Skills System (DBT-SS) in individuals with Intelligence Quotient 65-85 and recurrent self-harm. The study is primarily descriptive with 6 cases followed by repeated measurements (weekly; time series analysis). Primary outcome measure is frequency and severity of self-harming behavior, reported weekly 4 weeks before the start of the intervention, throughout the intervention and 12 weeks after the intervention has stopped.

DETAILED DESCRIPTION:
Not many psychotherapies are adapted to suit individuals with Intelligence Quotient(IQ) in the lower normal range. For individuals diagnosed with cognitive disability and self-harm, psychiatric treatment as usual often consists of only supportive meetings and sometimes heavy medication.

Dialectical Behavior therapy (DBT) is one of the evidence based treatments for individuals with self-harm and Borderline Personality Disorder. It is a comprehensive, multi component treatment, usually lasting a year or more. When offering DBT to individuals with cognitive disabilities or IQ in the lower normal range, it is necessary to alter the individual therapy procedures and skills group materials, while remaining adherent to DBT principles.

The Skills System is an adaptation of the standard DBT skills for individuals with cognitive challenges, well suited for IQ 65-85. When adapted DBT individual therapy integrates the Skills System as the skill group curriculum the treatment is called DBT-Skills System (DBT-SS). DBT-SS comprises weekly individual sessions, weekly group education and separate education for caregivers and/or near standing persons. The method is tested with positive effects on problem behaviors, however results need to be reproduced, and further tested in a randomized controlled trial. The handouts from Skills System has recently been translated to Swedish.

The current study aims to investigate the effect of Skills system on individuals with self-harm, IQ 65-85 and three or more symptoms of borderline personality disorder. A single-case time series design will be used with repeated, weekly measurements before, during and after the intervention is provided. 6 participants will be recruited in a pilot study, to investigate the feasibility of the method in a Swedish setting. Main outcome measures are frequency and severity of self-harming and aggressive behaviors, number of days with hospital admission and coercive care, number of medications, and self-rated level of daily functioning. Participation will last 64-70 weeks depending on when the group therapy starts in relation to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Ongoing contact with adult psychiatric clinic
* Intelligence Quotient 65-85
* Current self-harming behaviour at least twice the last six months
* Staff from residential care or near standing persons are able to participate in the treatment by participating in group sessions.

Exclusion Criteria:

* Schizophrenia or Bipolar illness type 1
* Substance abuse
* Non-psychiatric disorder significantly contributing to symptoms.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-12-10 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Deliberate self-harm | Baseline - 64 weeks
  Frequency of deliberate self-harm

SECONDARY OUTCOMES:
Problem behaviors | Baseline - 64 weeks
  Frequency of problem behaviors
Out-of control behavior | Baseline - 64 weeks
  Number of hours per week with out-of control behavior
Upset | Baseline - 64 weeks
  Number of hours per week when the individual is upset
Worried | Baseline - 64 weeks
  Number of hours per week when the individual is worried
Medication on demand | Baseline - 64 weeks
  Frequency of occasions with medication on demand
Visits to psychiatric emergency ward | Baseline - 64 weeks
  Frequency of visits to psychiatric emergency ward
Admission to hospital | Baseline - 64 weeks
  Number of days admitted to hospital
Coercive care | Baseline - 64 weeks
  Number of days with coercive care
Coercive acts | Baseline - 64 weeks
  Number of coercive acts
Psychotropic medications | Baseline - 64 weeks
  Number of psychotropic medications
Level of risk | Baseline - 64 weeks
  Measurement with Short-Term Assessment of Risk and Treatability
Resilience | Baseline - 64 weeks
  Measurement with Short-Term Assessment of Risk and Treatability
Vulnerability | Baseline - 64 weeks
  Measurement with Short-Term Assessment of Risk and Treatability
Level of functioning | Baseline - 64 weeks
  Self-rated by interview level of functioning in daily life with WHODAS 2.0

CONTACTS AND LOCATIONS:
Overall Officials: Sofie Westling, MD, PhD, Principal Investigator — Lund University
Locations (1):
- Division of Psychiatry, Region Skåne, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided